CLINICAL TRIAL: NCT02877849
Title: Brain Functional Connectivity During Early Recovery in Alcohol Use Disorder as a Marker for Relapse
Brief Title: Brain Functional Connectivity in Alcohol Use Disorder
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1606M89781
Record Dates: First submitted 2016-07-15; First posted 2016-08-24 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Alcohol Use Disorder
Keywords: fMRI; brain networks; biomarker; relapse; alcohol
MeSH Terms: conditions — Alcoholism; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals with Alcohol Use Disorder: Individuals with Alcohol Use Disorder will be recruited from Lodging Plus treatment program (Fairview Riverside Hospital, Minneapolis, MN). All patients will have between 2-3 weeks of abstinence from alcohol use. We will collect brain imaging data, this is an observational study.
  Interventions: Device: MRI: Brain Imaging data collection
- Healthy Volunteers: Healthy volunteers with comparable age and gender to the patient group will be recruited through community advertisements. We will collect brain imaging data, this is an observational study.
  Interventions: Device: MRI: Brain Imaging data collection

INTERVENTIONS:
Device: MRI: Brain Imaging data collection — This study has no intervention, it is observational. We will collect brain imaging data and behavioral assessments.

SUMMARY:
Due to the relapsing nature of alcoholism, excessive alcohol consumption represents a significant cost to US society ($249 billion in 20101). About 64% of those entering treatment will relapse within one year. New interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem. Using resting functional magnetic resonance imaging (fMRI) we have identified brain biomarkers that support long-term abstinence and brain biomarkers that predict relapse. Our data point to specific brain biomarkers that index higher relapse vulnerability at 11 weeks of abstinence. Many individuals, however, have already relapsed by this time. It is unknown whether these biomarkers can be identified earlier during the recovery period. We need to investigate whether this biomarker of relapse vulnerability can be identified during earlier stages of abstinence. Earlier identification of this biomarker will give valuable information for timely targeted interventions (e.g. closer monitoring, longer stay in treatment program, neuromodulation), increasing the chances of maintaining abstinence. The overall objective of this study is to identify biomarkers of relapse during early abstinence (2-3 weeks of abstinence). A secondary objective is to evaluate whether non-imaging measures such as craving6 and executive function7 add value to prediction models. Findings from this proposal will provide insight into the neurobiology of relapse vulnerability that will inform new treatment strategies needed to improve treatment outcome.

DETAILED DESCRIPTION:
BACKGROUND:

Due to the relapsing nature of alcoholism, excessive alcohol consumption represents a significant cost to US society ($249 billion in 2010). About 64% of those entering treatment will relapse within one year. Development of new and improved treatments that could be personalized to maximize the chance of maintaining abstinence in the first year will require advancement in understanding the behavioral and neural mechanisms underlying vulnerability to relapse during early abstinence. New interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem. Using resting functional magnetic resonance imaging (fMRI) we have identified brain biomarkers that support long-term abstinence and brain biomarkers that predict relapse. Our cross-sectional and longitudinal findings provide evidence that higher functional connectivity (FC), particularly between nucleus accumbens (NAcc) and dorsolateral prefrontal cortex (DLPFC) is a potential brain biomarker that supports abstinence. Resting NAcc-DLPFC FC is graded depending on abstinence length, with higher FC in long-term abstinent alcoholics (7 years of abstinence) than controls and intermediate FC in short-term abstinent alcoholics (11 weeks of abstinence). Further, lower NAcc-DLPFC FC at 11-weeks of abstinence can be a predictor of subsequent relapse (with 74% accuracy). Our data point to specific brain biomarkers that index higher relapse vulnerability at 11 weeks of abstinence. Many individuals, however, have already relapsed by this time and were not included in the studies above. It is unknown whether these biomarkers can be identified earlier during the recovery period. We need to investigate whether this biomarker of relapse vulnerability can be identified during earlier stages of abstinence. Earlier identification of this biomarker will give valuable information for timely targeted interventions (e.g. closer monitoring, longer stay in treatment program, neuromodulation), increasing the chances of maintaining abstinence.

PURPOSE OF THE STUDY:

Our long-term goal is to use identified brain and behavioral biomarkers to facilitate the development of new, personalized treatments that will support enduring abstinence in addiction. The overall objective of this study is to identify biomarkers of relapse during early abstinence (2-3 weeks of abstinence). A secondary objective is to evaluate whether non-imaging measures such as craving and executive function add value to prediction models. Findings from this study will provide insight into the neurobiology of relapse vulnerability that will inform new treatment strategies needed to improve treatment outcome.

SPECIFIC AIMS:

SA 1: To evaluate prediction accuracy of FC measures in individuals with alcohol use disorder (AUD) during early (2-3 weeks) abstinence. To evaluate whether non-imaging measures (e.g. craving, executive function) add value to FC prediction models we will test prediction models using (i) only imaging variables (FC during task and rest fMRI), (ii) only non-imaging variables, and (iii) a combination of imaging and non-imaging variables as predictors of time to relapse. Hypothesis: Based on compensatory mechanisms hypothesis, we expect that subsequent abstainers will have stronger NAcc-DLPFC FC when compared to subsequent relapsers and controls. Pilot data suggests that a combination of imaging and non-imaging variables will have high prediction accuracy. SA 2. To expand our examination of NAcc-DLPFC FC beyond resting state we will use the Reversal Learning (RL) task, which involves executive functioning and reward processing. Hypothesis: Pilot data suggests that subsequent abstainers will show higher task-related NAcc FC than relapsers and controls. Exploratory Aim: We will explore whether the strength of resting NAcc-DLPFC FC changes after performing the RL task. We will collect rest fMRI data before and after RL task performance in the scanner. Hypothesis: Based on previous findings of increased task-evoked activity in these regions, we hypothesize that patients will show increased resting NAcc-DLPFC FC after performing the RL task.

SIGNIFICANCE:

Addiction treatment outcomes are poor. Alcohol use disorder (AUD) in the U.S. remains an important public health problem with an estimated total annual cost to society of $249.5 billion. The chronic and relapsing nature of AUD is a major obstacle to successful recovery. We lack tools to subtype in alcohol use disorder (AUD). Subtyping in clinical populations can be an effective approach to model targeted interventions. For example, targeted treatment for breast cancer patients based on individual tumor estrogen receptor typing (biomarker) has improved outcomes from a 25 to 77% survival rate; there has not been a similar improvement in outcome for AUD treatment. We need to identify biomarkers in AUD that predict relapse and guide the development and selection of treatment based on subtypes to increase the chances of achieving long-term abstinence.

ELIGIBILITY:
Alcohol Use Disorder

INCLUSION CRITERIA:

* Age 18-60
* Ability to provide written consent and comply with study procedures
* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for Alcohol Use Disorder
* May have current comorbid drug use, but primary substance use disorder diagnosis needs to be based on alcohol use
* Must be enrolled in Lodging Plus (Fairview Riverside) treatment program
* Must have the intention to remain in program until the end of the study

EXCLUSION CRITERIA:

* Any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness>30 min, HIV)
* Any MRI scanning contraindications (i.e., metal implants, pacemakers, etc.)
* DSM-V criteria for psychiatric disorder, may have a lifetime but not current diagnosis of depression
* Primary current substance use disorder diagnosis on a substance other than alcohol except for caffeine or nicotine
* Clinical evidence for Wernicke-Korsakoff syndrome

Healthy controls

INCLUSION CRITERIA:

* Age 18-60
* Ability to provide written consent and comply with study procedures

EXCLUSION CRITERIA:

* Any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness>30 min, HIV)
* Any MRI scanning contraindications (i.e., metal implants, pacemakers, etc.)
* DSM-V criteria for psychiatric disorder, may have a lifetime but not current diagnosis of depression
* Primary current substance use disorder diagnosis on any substance such as alcohol, stimulant, opioids, etc. except for caffeine or nicotine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with alcohol use disorder will be only recruited from the Lodging Plus treatment program at Fairview Riverside in Minneapolis, MN Healthy volunteers will be recruited through community advertisements in Minneapolis, MN
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Brain connectivity measures at baseline | 2 years
  Brain imaging data will be collected using a 3T MRI scanner from both groups

SECONDARY OUTCOMES:
Follow-up abstinence status | 6 months after baseline assessments
  Subjects will be called back for follow-up brain imaging data collection, Timeline Follow-back to measure alcohol use, and relapse (abstinence vs relapse) status

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
As requested